CLINICAL TRIAL: NCT03551418
Title: Learning by Repetitive Viewing of Peer Modeling Patient Education Videos by Adults With Down Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interruption of COVID 19 pandemic
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AHC IRB 6884
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Down Syndrome; Trisomy 21
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repetitive video watching (Experimental): Repetitively watching a video of an adult with Down Syndrome washing his hands
  Interventions: Behavioral: Watching a video

INTERVENTIONS:
Behavioral: Watching a video — Watching a video of an adult with DS washing his hands

SUMMARY:
The learning of appropriate hand washing technique through repetitive watching of a video depicting an adult with DS washing his hands will be studied.

DETAILED DESCRIPTION:
This study is a next step in evaluating the use of videos depicting a person with DS demonstrating hand washing. The initial study demonstrated improvement in hand washing technique with a verbal explanation of hand washing technique using an Illinois Department of Public Health handout and viewing one of the handwashing videos one time. The study demonstrated a statistical significant difference between learning by viewing the handout and a video of an adult with DS washing his hands vs just viewing the handout.viewing a handout Likely due to small sample size, the study did not demonstrate statistical significance between watching the video of a person with DS washing his hands vs watching the other videos but the trend for the best improvement in handwashing technique was for the group viewing another person with DS demonstrating the handwashing. The hypothesis of this study is that repeated viewing of a video and practicing hand washing will lead to even greater improvement in hand washing technique.

ELIGIBILITY:
Inclusion criteria

Individuals with:

* DS aged 18 and older
* The ability to use a checklist or to be taught how to use a checklist
* The ability to use a tablet or to be taught how to use a tablet
* Access to an Internet connection

Exclusion criteria

Individuals who:

* Are not yet adults
* Are unwilling to consent and/or assent
* Are unable or unwilling to return the ADSC for the 1 month and 2 months follow up visits
* sensitivity to soap

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-09 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-08-16 (Actual)

PRIMARY OUTCOMES:
Appropriate hand washing technique | 2 months
  Measuring appropriate replicating of standard hand washing technique using a standard check list

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chicoine, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Adult Down Syndrome Center / Russell Institute for Research and Innovation, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No